CLINICAL TRIAL: NCT00702091
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Ramipril 10 mg Capsules Under Fasting Conditions
Brief Title: Bioequivalency Study of Ramipril 10 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, DRA-MA, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAMI-C10-PVFS-1
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ramipril — 10 mg capsule

SUMMARY:
The objective of this study was to prove the bioequivalence of Ramipril 10 mg capsules under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to Ramipril or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2005-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, two-period, 7 day washout

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Freeland, D.O., Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States